CLINICAL TRIAL: NCT04823065
Title: 4FMFES Positron Emission Tomography (PET) for Detection of Newly-diagnosed ER+ Endometrial and Ovarian Cancers
Brief Title: 4FMFES-PET Imaging of Endometrial and Ovarian Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, Head of clinical research, CRCHUS, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CIMS-2019-01
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Cancer; Ovarian Cancer
Keywords: PET; 4FMFES; Endometrial cancer; Ovarian cancer
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms | interventions — Loperamide; Butylscopolammonium Bromide

STUDY DESIGN:
Intervention Model Description: All recruited patients will undergo a 4FMFES-PET after biopsy confirmation of a ER+ endometrial cancer or suspicion of ovarian cancer. All patients are scanned prior to surgery.
  Patients are then randomly distributed for 3 different interventions aiming to reduce the intestinal peristalsis in order to diminish abdominal background generated by 4FMFES radio-metabolites.
  1. Control group: no intervention other than standard 4FMFES injection;
  2. 4 mg loperamide, per os, 15 minutes prior to 4FMFES injection;
  3. Repeated i.v. injection of 20 mg hyoscine-N-butylbromide at 0, 20 and 40 minutes after 4FMFES injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): 4FMFES injection is performed as usual, no supplemental medication is used.
- Loperamide (Experimental): Patients will receive 4 mg loperamide per os 15 minutes prior injection of the 4FMFES radiotracer dose. As a peristalsis inhibitor, it is expected that this medication will slow down the intestinal progression of the radio-metabolite bolus and thus spare the lower abdomen (where the assessed organs of interest are) of overwhelming background that could impair diagnosis.
  Interventions: Drug: Loperamide Pill
- Hyoscine-N-butylbromide (Experimental): In a similar fashion that what is used for some gastro-intestinal radiological examinations, repeated intravenous injection of 20 mg hyoscine-N-butylbromide will be applied at 0, 20 and 40 minutes following 4FMFES injection. As a peristalsis inhibitor, it is expected that this medication will slow down the intestinal progression of the radio-metabolite bolus and thus spare the lower abdomen (where the assessed organs of interest are) of overwhelming background that could impair diagnosis.
  Interventions: Drug: hyoscine-n-butylbromide

INTERVENTIONS:
Drug: Loperamide Pill — 4 mg Imodium, per os
  Other Names: Imodium
  Arms: Loperamide
Drug: hyoscine-n-butylbromide — 3 X 20 mg Buscopan, intravenous
  Other Names: Buscopan
  Arms: Hyoscine-N-butylbromide

SUMMARY:
This project is about exploring a novel method to detect ovarian and uterine cancers earlier and better. More precisely, a high-performance radioactive estrogen analog will be used to visualize hormone-sensitive uterine and ovarian tumors using PET imaging. Not only this imaging methodology could improve the whole-body assessment of those diseases, but will also hint clinicians about the optimal course of therapy to undertake.

The lead investigator's team designed in the past years an innovative radioactive estrogen derivative tracer (4FMFES) for the medical imaging modality termed Positron Emission Tomography (PET). The compound was first shown to be safe for human use. Recently, a clinical trial demonstrated that 4FMFES-PET is superior to any existing comparable tracer for detection of hormone-sensitive breast cancer patients. 4FMFES is particularly useful to pinpoint unsuspected metastases early, which allowed better breast cancer patient management and staging. 4FMFES and standard FDG PET imaging were shown to be complementary in breast cancer, the use of both techniques together providing a detection rate nearing 100%. Since ovarian and uterine cancers are about as likely to be targeted by 4FMFES as breast cancer, the use of this novel precision imaging method will be adapted to those other indications.

In general, the sooner a cancer is diagnosed and treated, the better the outcome of a patient will be. Gynecological cancers lack precise screening and detection tools. In particular, while a majority of uterine cancers are relatively well managed, patients burdened with metastatic burden have a much worse prognosis, and precise and early detection of those lesions will greatly help clinicians to better treat those complicated cases. As for ovarian cancers, they are usually devoid of clinical symptoms until late onset, which partly explain the high mortality rate of this disease. Hence, for both diseases, a precision, whole-body imaging technique will allow earlier assessment, followed by earlier intervention, resulting in improved survival rate and better quality of life for patients.

DETAILED DESCRIPTION:
Knowledge of estrogen receptor (ER) status is of paramount importance for breast cancer management. Mounting evidence supports an equally important role of ER status for uterine and ovarian cancers. Indeed, this prognostic factor was shown to stratify survival and progression-free rates, and to predict efficacy of ER-targeting adjuvant hormone therapy in those cancers. Between 70 and 80% of gynecological cancers expresses ER, akin to what is found in breast cancer. However, ER status is assessed by biopsy and hence is limited to primary lesions and to known, accessible metastases.

Commonly used diagnostic tools for gynecological cancers includes anatomical imaging modalities, such as echography, computed tomography (CT) and magnetic resonance imaging (MRI), with an increased role for metabolic [18F]-fluorodeoxyglucose positron emission tomography (FDG-PET) imaging, all yielding suboptimal tumor detection rate and poor specificity. Studies explored combination of FDG-PET/CT with [18F]-16α-fluoroestradiol (FES) PET/CT imaging to obtain whole-body assessment of ER status of both uterine and ovarian cancers, with FDG/FES uptake ratio correlating with grade and stage of disease. However, FES has many shortcomings, including rapid hepatic metabolism and binding to plasma globulins, resulting in a strong blood pool and in high nonspecific uptake, both detrimental to tumor detection.

The investigator's research center have designed a novel ER-targeting PET tracer, 4-fluoro-11β-methoxy-16α-[18F] fluoroestradiol (4FMFES) that addresses those flaws; 4FMFES is 2.5-fold more resistant to metabolism and does not bind to globulins. A phase II study comparing FES with 4FMFES-PET in breast cancer patients showed significantly reduced background with 4FMFES, resulting in improved tumor contrast and in an increased tumor detection rate. Preliminary results showed that addition of 4FMFES-PET to the standard FDG-PET allowed upstaging of ~20% of the breast cancer patients studied so far. Those breast cancer derived data forebode the potential of combined FDG- and 4FMFES-PET for whole-body diagnosis and ER status assessment for uterine and ovarian cancers.

Aim: Launch a phase I/II clinical trial evaluating the use of FDG and 4FMFES PET in ER+ uterine and ovarian cancer patients to enhance diagnostic confidence and accuracy, and to assess whole-body ER status non-invasively.

Specific aims:

1. Optimize imaging protocol for abdomen 4FMFES imaging: 4FMFES is eliminated by hepatobiliary excretion and as such generates strong signals in the intestinal tract, which could induce strong background and even false positives. Appropriate timing between 4FMFES injection and scan would allow optimal tumor uptake and minimal unwanted signal in the peritoneal area. Separately, pre-treatment with cholecystokinine (to pre-empty the gallbladder) or with opioids (to prevent intestinal peristalsis) will be explored as alternate ways of optimizing the protocol. A cohort of patients will be constituted in order to explore the best strategy to undertake for the rest of the study.
2. Evaluate the use of combined FDG and 4FMFES-PET for diagnosis and staging of ER+ uterine and ovarian cancers: Two cohorts of both uterine and ovarian cancer patients will be monitored by FDG and 4FMFES-PET/CT in sequence. Tumor uptake for each tracer will be compared. Number of detected lesion per patient using this protocol will be compared to whatever findings CT, or FDG alone would have found, and % of upstaged patients will be reported.
3. Correlate FDG and 4FMFES-PET tumor uptake with biopsy-derived grade and status: Every known, accessible lesion will be biopsied, and tumor grade and receptor status will be assessed. Correlation between pathological characteristics, and FDG and 4FMFES PET-derived tumor uptake will be drawn.

The lack of sensitive and accurate imaging tools for uterine and ovarian cancer means that diagnosis is too often achieved at late onset of those diseases. Not only the validation of 4FMFES-PET combined with standard FDG-PET should yield more precise, whole-body diagnostic and staging, but also could predict prognosis and targeted therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women who received a biopsy-confirmed diagnosis of a ER+ endometrial cancer, or;
* Women with a suspected ovarian cancer, or;
* Women with recurrent endometrial or ovarian cancer and with a ER+ primary tumor, and;
* Planned surgery, and;
* Stage 1A cancer and more, with primary more than 1 cm, and;
* Able to tolerate supine position, and;
* Written consent given by the patient.

Exclusion Criteria:

* Pregnancy, or;
* Replacement hormone therapy concomitant to 4FMFES-PET, or;
* Use of estrogen-based oral contraceptives concomitant to 4FMFES-PET, or;
* Anti-tumor hormone therapy that compete with estrogen receptors concomitant to 4FMFES-PET, such as tamoxifen and fulvestrant. Withdrawal of such therapies 8 weeks prior to the 4FMFES-PET scan will enable the patient to the imaging test, or;
* Cirrhosis, acute or chronic hepatitis, or any other hepatic problem that might impede the normal elimination of the PET tracer, or;
* Hypersentivity to either FDG or 4FMFES, or any of their consittuants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate 4FMFES-PET diagnostic properties in endometrial and ovarian cancers | 48 months
  4FMFES-PET ability to detect tumors and assess extend of the disease will be monitored with both qualitative and semi-quantitative parameters. The 4FMFES uptake of each assessed lesion will be reported as Standard Uptake Value (SUV).
Compare 4FMFES-PET with standard FDG-PET in gynaecological cancers. | 48 months
  When available, 4FMFES-PET sessions will be scheduled within 2 weeks of a standard FDG-PET examination. The Standard Uptake Value (SUV)-derived tumor uptake will be compared between each tracer. The radiological, surgical and pathological assessment will be used as standard confirmation of the presence and size of tumors to confirm PET's finding.
Use pharmaceutical intervention to slow down peristalsis to improve lower-abdomen 4FMFES-PET | 48 months
  Patients that undergoes 4FMFES-PET will be assigned to 1) no-intervention control group; 2) 4 mg loperamide per os; 3) repeated 20 mg hyoscine-N-butylbromide injection. The volume occupied by excreted radio-metabolites (via the hepatobiliary pathway) will be estimated by applying a SUV < 4.0 threshold on a region-of-interest covering the whole abdomen.

CONTACTS AND LOCATIONS:
Overall Officials: Éric Turcotte, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Paquette M, Espinosa-Bentancourt E, Lavallee E, Phoenix S, Lapointe-Milot K, Bessette P, Guerin B, Turcotte EE. 18F-4FMFES and 18F-FDG PET/CT in Estrogen Receptor-Positive Endometrial Carcinomas: Preliminary Report. J Nucl Med. 2022 May;63(5):702-707. doi: 10.2967/jnumed.121.262617. Epub 2021 Aug 19. PMID 34413142